CLINICAL TRIAL: NCT00957671
Title: Anterior Pituitary Hormone Replacement in Traumatic Brain Injury
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Collaborators: The Moody Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 03-034
Record Dates: First submitted 2009-08-10; First posted 2009-08-12 (Estimated); Results first posted 2018-05-15 (Actual); Last update posted 2018-06-29 (Actual); Status verified 2018-05

CONDITIONS: Growth Hormone Deficiency; Traumatic Brain Injury
Keywords: TBI; Traumatic Brain injury; Growth hormone deficiency; Anterior pituitary hormone; Recombinant human growth Hormone; Genotropin
MeSH Terms: conditions — Dwarfism, Pituitary; Brain Injuries, Traumatic | interventions — Growth Hormone; Human Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Human Growth Hormone (Experimental): recombinant human growth hormone (rhGH) self administered daily for one year
  Interventions: Drug: Recombinant human growth hormone

INTERVENTIONS:
Drug: Recombinant human growth hormone — 200 mcg daily for two months, followed by 400 mcg daily for two months followed by 600 mcg daily for term of treatment period (one year total)
  Other Names: Genotropin; Somatropin; hGH

SUMMARY:
Fifteen to twenty percent of adults who suffer a traumatic brain injury (TBI) that requires hospitalization and rehabilitation have been found to have growth hormone (GH) deficiency by GH stimulation testing. Moreover, abnormalities have also been established for the cortisol and thyroid axis. The hypothesis of this proposal is that hormone replacement in TBI patients with documented abnormalities in the GH, thyroid, or cortisol axis will improve muscle function, body composition, aerobic capacity (GH) and tests of neuropsychologic function (GH, thyroid, cortisol).

DETAILED DESCRIPTION:
This protocol is designed to screen and detect evidence of pituitary hormone deficiency in adults following traumatic brain injury. Growth hormone deficiency will be replaced for a period of one year. Subject will not be screened until at least one year following brain injury to allow for natural recovery of hormone function.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 21 and older.
* Documented moderate to severe traumatic brain injury at least one year post injury.

Exclusion Criteria:

* The only absolute exclusionary medication will be an anticoagulant (Coumadin) because of the risk of bleeding during the possible muscle biopsy procedure and daily injections of rhGH in the GH arm of the study.
* Any subject with a history of hepatitis or a 3-fold elevation of liver function tests (Alk phos, alanine aminotransferase (ALT), aspartate aminotransferase (AST)). We are uncertain of the effects of hormone replacement such as rhGH on the liver, so we will exclude any subjects with hepatitis. This exclusion applies only to subjects who would be enrolled in the GH arm of the study.
* Subjects who are deficient in cortisol or thyroid at screening will be excluded until hormone abnormalities have been corrected.
* Subjects with chronic pain who are being managed with narcotics will be excluded as the effects of central nervous system depressants may interfere with study test results.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2003-11; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Randall J Urban, M.D., Principal Investigator — The University of Texas Medical Branch at Galveston
Locations (2):
- United States (2):
  - Transitional Learning Center, Galveston, Texas
  - The University of Texas Medical Branch at Galveston, Galveston, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects with a history of mild to severe traumatic brain injury were recruited from 2010 to 2014. Subjects were screened for abnormal growth hormone secretion by glucagon stimulation test. 19 subjects were screened for this study. 15 of the subjects met final inclusion/exclusion criteria and began the treatment phase.
Groups:
- Human Growth Hormone: recombinant human growth hormone (rhGH) self administered daily for one year.
  Human Growth Hormone: 200 mcg daily for two months, followed by 400 mcg daily for two months followed by 600 mcg daily for term of treatment period (one year total).
Period: Overall Study
Arm/Group | Human Growth Hormone
Started | 15 (15 subjects began the treatment phase.)
Completed | 15 (15 subjects completed the treatment phase of the study.)
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 15 subjects with a history of mild to severe traumatic brain injury and abnormal growth hormone secretion were enrolled in this trial.
Groups:
- Human Growth Hormone: Recombinant human growth hormone (rhGH) self administered daily for one year
  Human Growth Hormone: 200 mcg daily for two months, followed by 400 mcg daily for two months followed by 600 mcg daily for term of treatment period (one year total)
Arm/Group | Human Growth Hormone
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.5 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 10
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15
Age at time of injury [Mean (Standard Deviation); unit: years] | 34.3 (15.7)

OUTCOME MEASURES:

1. Primary Outcome: Maximum Oxygen Uptake at Baseline.
Description: Maximum Oxygen Uptake was measured during cardiorespiratory testing using a modified Balke protocol with expired gases collected and analyzed by an automated metabolic cart.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: mL/kg/min
Arm/Group | Human Growth Hormone
Number analyzed (Participants) | 15
mL/kg/min | 29.0 (7.2)

2. Primary Outcome: Maximum Oxygen Uptake After One Year of Human Growth Hormone Replacement Therapy.
Description: as for outcome 1
Time Frame: one year
Measure: Mean (Standard Deviation); unit: mL/kg/min
Arm/Group | Human Growth Hormone
Number analyzed (Participants) | 15
mL/kg/min | 32.1 (7.4)

3. Primary Outcome: Minute Ventilation at Baseline.
Description: Minute ventilation was measured during cardiorespiratory testing using a modified Balke protocol with expired gases collected and analyzed by an automated metabolic cart.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: L/minute
Arm/Group | Human Growth Hormone
Number analyzed (Participants) | 15
L/minute | 90.4 (24.2)

4. Primary Outcome: Minute Ventilation After One Year of Human Growth Hormone Replacement Therapy.
Description: as for outcome 3
Time Frame: one year
Measure: Mean (Standard Deviation); unit: L/minute
Arm/Group | Human Growth Hormone
Number analyzed (Participants) | 15
L/minute | 102.4 (23.1)

5. Primary Outcome: Respiratory Exchange Ratio at Baseline.
Description: Respiratory exchange ratio was measured during cardiorespiratory testing using a modified Balke protocol with expired gases collected and analyzed by an automated metabolic cart.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: ratio of CO2/O2
Arm/Group | Human Growth Hormone
Number analyzed (Participants) | 15
ratio of CO2/O2 | 1.27 (0.12)

6. Primary Outcome: Respiratory Exchange Ratio After One Year of Human Growth Hormone Replacement Therapy.
Description: as for outcome 5
Time Frame: one year
Measure: Mean (Standard Deviation); unit: ratio of CO2/O2
Arm/Group | Human Growth Hormone
Number analyzed (Participants) | 15
ratio of CO2/O2 | 1.27 (0.10)

7. Primary Outcome: Oxygen Pulse at Baseline.
Description: Oxygen Pulse was measured during cardiorespiratory testing using a modified Balke protocol with expired gases collected and analyzed by an automated metabolic cart. Oxygen pulse is calculated by dividing VO2 consumed (mL/min) by heart rate (beats/min) yielding mL/beat. This provides an estimate of cardiac stroke volume.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: mL/beat
Arm/Group | Human Growth Hormone
Number analyzed (Participants) | 15
mL/beat | 15.2 (4.1)

8. Primary Outcome: Oxygen Pulse After One Year of Human Growth Hormone Replacement Therapy.
Description: as for outcome 7
Time Frame: one year
Measure: Mean (Standard Deviation); unit: mL/beat
Arm/Group | Human Growth Hormone
Number analyzed (Participants) | 15
mL/beat | 16.4 (4.2)

9. Secondary Outcome: Neuropsychological Function as Measured by California Verbal Learning Test-II With Total Recall at Baseline.
Description: The California Verbal Learning Test II (CVLT-II) is a comprehensive assessment of verbal learning and memory. Subjects are read a list of 16 words. Total recall is a sum of all word list items correctly recalled immediately on learning trials 1 through 5. Data is reported as raw scores. Score range is 0 (lowest) to 80 (highest). A higher score indicates a better outcome.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Human Growth Hormone
Number analyzed (Participants) | 15
scores on a scale | 45.7 (10.8)

10. Secondary Outcome: Neuropsychological Function as Measured by California Verbal Learning Test-II With Total Recall After 1 Year of Human Growth Hormone Replacement Therapy.
Description: as for outcome 9
Time Frame: One year
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Human Growth Hormone
Number analyzed (Participants) | 15
scores on a scale | 51.0 (9.4)

11. Secondary Outcome: Neuropsychological Function as Measured by California Verbal Learning Test-II With Delayed Recall at Baseline.
Description: The California Verbal Learning Test II (CVLT-II) is a comprehensive assessment of verbal learning and memory. Subjects are read a list of 16 words. Delayed recall is a sum of all word list items correctly recalled after a 25 minute delay on learning trials 1 through 5. Data is reported as raw scores. Score range is 0 (lowest) to 80 (highest). A higher score indicates a better outcome.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Human Growth Hormone
Number analyzed (Participants) | 15
scores on a scale | 9.9 (3.8)

12. Secondary Outcome: Neuropsychological Function as Measured by California Verbal Learning Test-II With Delayed Recall After 1 Year of Human Growth Hormone Replacement Therapy.
Description: as for outcome 11
Time Frame: One year
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Human Growth Hormone
Number analyzed (Participants) | 15
scores on a scale | 11.2 (2.6)

13. Secondary Outcome: Neuropsychological Function as Measured by Brief Visuospatial Memory Test-R With Total Recall at Baseline
Description: The Brief Visuospatial Memory Test is measure of visual memory. The subject views a stimulus page with 6 shapes on it for 10 seconds. The subjects are then asked to draw as many figures as they remember in the correct locations as possible. Total recall is a measure of the subjects memory immediately after viewing the stimulus page. Data is reported as raw scores. Scores range from 0 (lowest) to 36 (highest). A higher score indicates a better outcome.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Human Growth Hormone
Number analyzed (Participants) | 15
scores on a scale | 18.7 (5.7)

14. Secondary Outcome: Neuropsychological Function as Measured by Brief Visuospatial Memory Test-R With Total Recall After 1 Year of Human Growth Hormone Replacement Therapy.
Description: as for outcome 13
Time Frame: one year
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Human Growth Hormone
Number analyzed (Participants) | 15
scores on a scale | 22.7 (5.1)

15. Secondary Outcome: Neuropsychological Function as Measured by Brief Visuospatial Memory Test-R With Delayed Recall at Baseline
Description: The Brief Visuospatial Memory Test is measure of visual memory. The subject views a stimulus page with 6 shapes on it for 10 seconds. The subjects are then asked to draw as many figures as they remember in the correct locations as possible. The delayed recall is a measure of the subjects memory after a 25 minutes delay. The participants are asked to freely recall and again draw the six figures.Data is reported as raw scores. Scores range from 0 (lowest) to 36 (highest). A higher score indicates a better outcome.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Human Growth Hormone
Number analyzed (Participants) | 15
scores on a scale | 7.2 (2.9)

16. Secondary Outcome: Neuropsychological Function as Measured by Brief Visuospatial Memory Test-R With Delayed Recall After 1 Year of Human Growth Hormone Replacement Therapy
Description: as for outcome 15
Time Frame: one year
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Human Growth Hormone
Number analyzed (Participants) | 15
scores on a scale | 9.1 (2.2)

17. Secondary Outcome: Neuropsychological Function as Measured by Digit Span Total at Baseline
Description: Digit Span; Wechsler Memory Scale III (WMS III).
  Digits Forward is a test of digit span (range = 3 to 9 digits) consisting of seven items (each with 2 trials). Digits Backward is a test of digit span (range = 3 to 9 digits); however the participant must provide the presented sequence in reverse order. The test consists of seven items (each with 2 trials). Total score is calculated by adding the scores from forward and backward. Data is reported as raw scores. Score ranges are 0 (lowest) to 32 (highest). A higher score indicates a better outcome.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Human Growth Hormone
Number analyzed (Participants) | 15
scores on a scale | 16.0 (4.5)

18. Secondary Outcome: Neuropsychological Function as Measured by Digit Span Total After One Year of Human Growth Hormone Replacement Therapy.
Description: as for outcome 17
Time Frame: one year
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Human Growth Hormone
Number analyzed (Participants) | 15
scores on a scale | 17.0 (3.9)

19. Secondary Outcome: Neuropsychological Function as Measured by Processing Speed Index at Baseline
Description: Processing Speed Index is a subcategory of the Wechsler Adult Intelligence Scale III (WAIS-III). Processing speed refers to the speed of cognitive processes and response output.
  This index is comprised of performances on two separate tests of visuomotor speed of information processing ability. On one test (Coding) participants refer to a key on top of a page to translate non-verbal symbols to an alpha-numeric digit. The participants then fill in boxes with the correct symbol assigned to a particular number. On the other test (Symbol Search) participants are asked to visually scan and mark items that are identical to one of two targets. If neither target is shown in the array the participant must mark out the work "NO". Total correct responses for both task within 120 seconds are recorded.
  Ranges are 0 (lowest) to 150 (highest) with 100 being the normal average. A higher score indicates a better outcome.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Human Growth Hormone
Number analyzed (Participants) | 15
scores on a scale | 102.3 (14.9)

20. Secondary Outcome: Neuropsychological Function as Measured by Processing Speed Index After One Year of Human Growth Hormone Replacement Therapy.
Description: as for outcome 19
Time Frame: one year
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Human Growth Hormone
Number analyzed (Participants) | 15
scores on a scale | 106.6 (15.0)

21. Secondary Outcome: Neuropsychological Function as Measured by Letter Fluency at Baseline
Description: Letter Fluency is a condition measured as part of the subcategory, Verbal Fluency, in the Delis-Kaplan Executive Function System (D-KEFS). Subjects are asked to name as many words as they can starting with a specified letter for 60 seconds. The words can not be names, places, numbers or grammatical variants of previous answers. Repeated answers are not scored as a correct response. There are 3 trials, with 3 different letters. The total number of correct responses is totaled for all 3 trials and a Letter Fluency Score is given. A higher score is considered better. There is no set range as the score depends on how many correct words the subject relays in the given time period.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Human Growth Hormone
Number analyzed (Participants) | 15
scores on a scale | 38.5 (14.5)

22. Secondary Outcome: Neuropsychological Function as Measured by Letter Fluency After One Year of Human Growth Hormone Replacement Therapy
Description: as for outcome 21
Time Frame: one year
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Human Growth Hormone
Number analyzed (Participants) | 15
scores on a scale | 35.4 (13.0)

23. Secondary Outcome: Depression as Measured by the Beck Depression Inventory at Baseline.
Description: Beck Depression Inventory (BDI-II) is used to measure the severity of depression symptoms. The BDI-II contains 21 questions, each answer being scored on a scale value of 0 to 3. Higher total scores indicate more severe depressive symptoms. The standardized cutoffs are: 0-13: minimal depression; 14-19: mild; depression; 20-28: moderate depression; 29-63: severe depression.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Human Growth Hormone
Number analyzed (Participants) | 15
scores on a scale | 13.8 (9.7)

24. Secondary Outcome: Depression as Measured by Beck Depression Inventory After One Year of Human Growth Hormone Replacement Therapy.
Description: as for outcome 23
Time Frame: one year
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Human Growth Hormone
Number analyzed (Participants) | 15
scores on a scale | 6.2 (6.9)

25. Secondary Outcome: Fatigue as Measured Using Fatigue Severity Scale at Baseline.
Description: Fatigue Severity Scale (FSS) is a measure of fatigue and how that fatigue interferes with life. It is a 9-item scale, with a range from 9 to 63, with a higher number indicating greater severity.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Human Growth Hormone
Number analyzed (Participants) | 15
scores on a scale | 44.3 (13.5)

26. Secondary Outcome: Fatigue Measured Using the Fatigue Severity Scale After One Year of Human Growth Hormone Therapy.
Description: as for outcome 25
Time Frame: one year
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Human Growth Hormone
Number analyzed (Participants) | 15
scores on a scale | 34.0 (12.5)

27. Secondary Outcome: Muscle Function in Male Subjects Measured Using Maximum Isometric Leg Extension by Biodex Pro 4 at Baseline.
Description: Maximum torque production during isometric contraction of the knee extensor muscles.
Time Frame: baseline
Population: This is the data for the 10 male subjects enrolled in this study.
Measure: Mean (Standard Deviation); unit: Newton-Meters
Arm/Group | Human Growth Hormone
Number analyzed (Participants) | 10
Newton-Meters | 206.0 (32.41)

28. Secondary Outcome: Muscle Function in Male Subjects Measured Using Maximum Isometric Leg Extension by Biodex Pro 4 After One Year of Human Growth Hormone Replacement Therapy.
Description: Maximum torque production during isometric contraction of the knee extensor muscles.
Time Frame: one year
Population: This is the data for the 10 male subjects in this study.
Measure: Mean (Standard Deviation); unit: Newton-Meters
Arm/Group | Human Growth Hormone
Number analyzed (Participants) | 10
Newton-Meters | 209.6 (37.65)

29. Secondary Outcome: Muscle Function in Male Subjects Measured Using Maximum Isokinetic Leg Extension by Biodex Pro 4 at Baseline.
Description: Maximum torque production during maximal isokinetic contractions at 90 degrees per second.
Time Frame: baseline
Population: This data is for the 10 male subjects enrolled in this study.
Measure: Mean (Standard Deviation); unit: Newton-Meters
Arm/Group | Human Growth Hormone
Number analyzed (Participants) | 10
Newton-Meters | 175.2 (36.61)

30. Secondary Outcome: Muscle Function in Male Subjects Measured Using Maximum Isokinetic Leg Extension by Biodex Pro 4 After One Year of Human Growth Hormone Replacement Therapy.
Description: Maximum torque production during maximal isokinetic contractions at 90 degrees per second.
Time Frame: one year
Population: This data is for the 10 male subjects in this study.
Measure: Mean (Standard Deviation); unit: Newton-Meters
Arm/Group | Human Growth Hormone
Number analyzed (Participants) | 10
Newton-Meters | 182.6 (45.29)

31. Secondary Outcome: Muscle Fatigue as Measured by Biodex Pro 4 at Baseline.
Description: Muscle fatigue is measured using repetitive isokinetic contractions of the knee extensors at 90 degrees per second. Each subject was asked to produce 40 contractions at full force. Data is presented as % of maximum torque at the 40th contraction in the fatigue protocol.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: Percent of Maximum Torque
Arm/Group | Human Growth Hormone
Number analyzed (Participants) | 15
Percent of Maximum Torque | 35.1 (6.30)

32. Secondary Outcome: Muscle Fatigue as Measured by Biodex Pro 4 After One Year of Human Growth Hormone Replacement Therapy.
Description: as for outcome 31
Time Frame: one year
Measure: Mean (Standard Deviation); unit: Percent of Maximum Torque
Arm/Group | Human Growth Hormone
Number analyzed (Participants) | 15
Percent of Maximum Torque | 36.9 (9.89)

33. Secondary Outcome: Body Mass in Male Subjects as Measured by Dual Energy X-Ray Absorptiometry (DEXA) at Baseline.
Description: Body mass was calculated from whole body scan taken using a GE Lunar iDEXA.
Time Frame: baseline
Population: This data is for the 10 male subjects in the study.
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Human Growth Hormone
Number analyzed (Participants) | 10
kilograms | 96.04 (18.38)

34. Secondary Outcome: Body Mass in Male Subjects as Measured by Dual Energy X-Ray Absorptiometry (DEXA) After One Year of Human Growth Hormone Replacement Therapy.
Description: Body mass was calculated from whole body scan taken using a GE Lunar iDEXA
Time Frame: one year
Population: This is the data for the 10 male subjects in the study.
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Human Growth Hormone
Number analyzed (Participants) | 10
kilograms | 96.55 (19.67)

35. Secondary Outcome: Lean Body Mass in Male Subjects as Measured by Dual Energy X-Ray Absorptiometry (DEXA) at Baseline
Description: Lean Body mass was calculated from whole body scan taken using a GE Lunar iDEXA
Time Frame: baseline
Population: This data is for the 10 male subjects enrolled in this study.
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Human Growth Hormone
Number analyzed (Participants) | 10
kilograms | 61.68 (7.55)

36. Secondary Outcome: Lean Body Mass in Male Subjects as Measured by Dual Energy X-Ray Absorptiometry (DEXA) After One Year of Human Growth Hormone Replacement Therapy.
Description: Lean Body mass was calculated from whole body scan taken using a GE Lunar iDEXA
Time Frame: one year
Population: This data is for the 10 male subjects enrolled in the study.
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Human Growth Hormone
Number analyzed (Participants) | 10
kilograms | 63.70 (8.14)

37. Secondary Outcome: Fat Free Mass in Male Subjects as Measured by Dual Energy X-Ray Absorptiometry (DEXA) at Baseline.
Description: Fat free mass is calculated from whole body scan measured using a GE Lunar iDEXA.
Time Frame: baseline
Population: This data is for the 10 male subjects enrolled in this study.
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Human Growth Hormone
Number analyzed (Participants) | 10
kilograms | 31.19 (13.75)

38. Secondary Outcome: Fat Free Mass in Male Subjects as Measured by Dual Energy X-Ray Absorptiometry (DEXA) After One Year of Human Growth Hormone Replacement Therapy.
Description: Fat free mass is calculated from whole body scan measured on a GE Lunar iDEXA.
Time Frame: one year
Population: This is the data for the 10 male subjects enrolled in the study.
Measure: Mean (Standard Deviation); unit: kilogram
Arm/Group | Human Growth Hormone
Number analyzed (Participants) | 10
kilogram | 29.67 (14.30)

39. Secondary Outcome: Percent Body Fat as Measured by Dual Energy X-Ray Absorptiometry (DEXA) at Baseline.
Description: Percent body fat is calculated from a whole body scan measured on a GE Lunar iDEXA.
Time Frame: baseline
Population: This data is for the 10 male subjects enrolled in this study.
Measure: Mean (Standard Deviation); unit: percent of body fat
Arm/Group | Human Growth Hormone
Number analyzed (Participants) | 10
percent of body fat | 32.47 (8.47)

40. Secondary Outcome: Percent Body Fat in Male Subjects as Measured by Dual Energy X-Ray Absorptiometry (DEXA) After One Year of Human Growth Hormone Replacement Therapy.
Description: Percent body fat is calculated from a whole body scan measured on a GE Lunar iDEXA.
Time Frame: one year
Population: This data is for the 10 male subjects in the study.
Measure: Mean (Standard Deviation); unit: percent of body fat
Arm/Group | Human Growth Hormone
Number analyzed (Participants) | 10
percent of body fat | 30.5 (9.40)

41. Secondary Outcome: Muscle Function in Female Subjects Measured Using Maximum Isometric Leg Extension by Biodex Pro 4 at Baseline.
Description: Maximum torque production during isometric contraction of the knee extensor muscles.
Time Frame: baseline
Population: This data is for the 5 female subjects enrolled in this study.
Measure: Mean (Standard Deviation); unit: Newton-Meters
Arm/Group | Human Growth Hormone
Number analyzed (Participants) | 5
Newton-Meters | 131.5 (26.38)

42. Secondary Outcome: Muscle Function in Female Subjects Measured Using Maximum Isometric Leg Extension by Biodex Pro 4 After One Year of Human Growth Hormone Replacement Therapy
Description: Maximum torque production during isometric contraction of the knee extensor muscles.
Time Frame: one year
Population: This data is for the 5 female subjects in the study.
Measure: Mean (Standard Deviation); unit: Newton-Meters
Arm/Group | Human Growth Hormone
Number analyzed (Participants) | 5
Newton-Meters | 130.7 (34.77)

43. Secondary Outcome: Muscle Function in Female Subjects Measured Using Maximum Isokinetic Leg Extension by Biodex Pro 4 at Baseline
Description: Maximum torque production during maximal isokinetic contractions at 90 degrees per second.
Time Frame: baseline
Population: This data is for the 5 female subjects enrolled in this study.
Measure: Mean (Standard Deviation); unit: Newton-Meters
Arm/Group | Human Growth Hormone
Number analyzed (Participants) | 5
Newton-Meters | 103.9 (12.56)

44. Secondary Outcome: Muscle Function in Female Subjects Measured Using Maximum Isokinetic Leg Extension by Biodex Pro 4 After One Year of Human Growth Hormone Replacement Therapy
Description: Maximum torque production during maximal isokinetic contractions at 90 degrees per second.
Time Frame: one year
Population: This data is for the 5 female subjects enrolled in this study.
Measure: Mean (Standard Deviation); unit: Newton-Meters
Arm/Group | Human Growth Hormone
Number analyzed (Participants) | 5
Newton-Meters | 99.6 (17.58)

45. Secondary Outcome: Perceptual Fatigability as Measured by a Fatigue Rating Scale at Baseline.
Description: Perceptual fatigue was measured before and directly after performing the muscle fatigue exercise protocol (40 continuous maximal force isokinetic knee extensions at 90 degress per second). Subjects were asked to rate their fatigue on a scale of 0-10 with 0 being no fatigue at all and 10 being extreme fatigue. Data is presented as change in fatigue rating induced by exercise testing.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Human Growth Hormone
Number analyzed (Participants) | 15
units on a scale | 3.78 (1.75)

46. Secondary Outcome: Perceptual Fatigability as Measured by a Fatigue Rating Scale After One Year of Human Growth Hormone Therapy.
Description: as for outcome 45
Time Frame: one year
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Human Growth Hormone
Number analyzed (Participants) | 15
units on a scale | 3.17 (1.54)

47. Secondary Outcome: Body Mass in Female Subjects as Measured by Dual Energy X-Ray Absorptiometry (DEXA) at Baseline.
Time Frame: baseline
Population: This is the data for the 5 females in the study.
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Human Growth Hormone
Number analyzed (Participants) | 5
kilograms | 75.64 (10.80)

48. Secondary Outcome: Body Mass in Female Subjects as Measured by Dual Energy X-Ray Absorptiometry (DEXA) After One Year of Human Growth Hormone Replacement Therapy
Description: Body mass was calculated from whole body scan taken using a GE Lunar iDEXA
Time Frame: one year
Population: This data represents the 5 females in the study.
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Human Growth Hormone
Number analyzed (Participants) | 5
kilograms | 76.54 (10.57)

49. Secondary Outcome: Lean Body Mass in Female Subjects as Measured by Dual Energy X-Ray Absorptiometry (DEXA) at Baseline
Description: Lean Body mass was calculated from whole body scan taken using a GE Lunar iDEXA.
Time Frame: baseline
Population: This data is for the 5 female subjects in the study.
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Human Growth Hormone
Number analyzed (Participants) | 5
kilograms | 43.84 (1.42)

50. Secondary Outcome: Lean Body Mass in Female Subjects as Measured by Dual Energy X-Ray Absorptiometry (DEXA) After One Year of Human Growth Hormone Replacement Therapy.
Description: Lean Body mass was calculated from whole body scan taken using a GE Lunar iDEXA
Time Frame: one year
Population: This data is for the 5 female subjects in the study.
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Human Growth Hormone
Number analyzed (Participants) | 5
kilograms | 44.92 (3.47)

51. Secondary Outcome: Fat Free Mass in Female Subjects as Measured by Dual Energy X-Ray Absorptiometry (DEXA) at Baseline.
Description: Fat free mass is calculated from whole body scan measured using a GE Lunar iDEXA.
Time Frame: baseline
Population: This data is for the 5 female subjects in the study.
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Human Growth Hormone
Number analyzed (Participants) | 5
kilograms | 29.31 (9.86)

52. Secondary Outcome: Fat Free Mass in Female Subjects as Measured by Dual Energy X-Ray Absorptiometry (DEXA) After One Year of Human Growth Hormone Replacement Therapy
Description: Fat free mass is calculated from whole body scan measured on a GE Lunar iDEXA.
Time Frame: one year
Population: This is the data for the 5 female subjects.
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Human Growth Hormone
Number analyzed (Participants) | 5
kilograms | 29.15 (8.74)

53. Secondary Outcome: Percent Body Fat in Female Subjects as Measured by Dual Energy X-Ray Absorptiometry (DEXA) at Baseline.
Description: Percent body fat is calculated from a whole body scan measured on a GE Lunar iDEXA.
Time Frame: baseline
Population: This data is for the 5 female subjects enrolled in the study.
Measure: Mean (Standard Deviation); unit: percent of body fat
Arm/Group | Human Growth Hormone
Number analyzed (Participants) | 5
percent of body fat | 38.92 (8.17)

54. Secondary Outcome: Percent Body Fat in Female Subjects as Measured by Dual Energy X-Ray Absorptiometry (DEXA) After One Year of Human Growth Hormone Replacement Therapy.
Description: Percent body fat is calculated from a whole body scan measured on a GE Lunar iDEXA.
Time Frame: one year
Population: This data is for the 5 female subjects enrolled in this study.
Measure: Mean (Standard Deviation); unit: percent of body fat
Arm/Group | Human Growth Hormone
Number analyzed (Participants) | 5
percent of body fat | 38.74 (6.84)

ADVERSE EVENTS:
Arm/Group | Human Growth Hormone
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No